CLINICAL TRIAL: NCT06197490
Title: Renal Impact of KAFTRIO in Mucoviscidose Population
Acronym: IRT-MUCO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5080; 69HCL23_1169 (Other: Easydore)
Record Dates: First submitted 2023-12-11; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; KAFTRIO; renal impact; lithiasis
MeSH Terms: conditions — Cystic Fibrosis; Lithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with cystic fibrosis, eligible for KAFTRIO therapy: Patient with cystic fibrosis, eligible for KATRIO, over 18 years old.
  Interventions: Biological: Evaluation of the parameters of the lithiasis assessment before and after KAFTRIO initiation; Drug: Collection of Arterial pressure, metabolic data, kidney function, proteinuria and hematuria before and after KATRIO initiation

INTERVENTIONS:
Biological: Evaluation of the parameters of the lithiasis assessment before and after KAFTRIO initiation — Collection of Uricuria, phosphaturie, calciuria, magnesuria, glycosuria, citraturia, oxaluria, before and after initiation of KAFTRIO
Drug: Collection of Arterial pressure, metabolic data, kidney function, proteinuria and hematuria before and after KATRIO initiation — Arterial pressure, glycemia, glycated hemoglobin, lipid profile, weight, serum and urinary electrolytes, hepatic check, complete blood count, calcium phosphate balance and urinary sediment analysis before and after initiation of KAFTRIO

SUMMARY:
The objective of this study is to describe the renal impact of Elexacaftor-Teacaftor-Ivacaftor, a triple modulator therapy of CFTR channel, in patients with cystic fibrosis. This new treatment acts on the CFTR channel, which is expressed at the level of the nephrons. The objective is to study the changes in plasma and urinary parameters, including metabolic explorations of urolithiasis, change in volemic parameters, renal function, urinary sediment and nutritional and glycemic parameters, in newly treated patients, through the data collected at introduction of the treatment and during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cystic fibrosis
* More than 18 years old
* Eligible for KAFTRIO

Exclusion Criteria:

* KAFTRIO contraindication
* Patient less than 18 years old
* Dialysis patient
* Pregnant woman
* Greffed patient
* Patient opposition to data collection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with cystic fibrosis followed at Centre Hospitalier Lyon Sud (in the reference and competence center for cystic fibrosis)
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Modification of the parameters of the lithiasis assessment | 1 month after initiation of KAFTRIO
  Change in blood phosphorus and calcium metabolism ; Change in calciuria mmol/d ;Change in urinary pH, urinary specific gravity (g/mL) and crystalluria
Modification of the parameters of the lithiasis assessment | 7 months after initiation of KAFTRIO
  Change in blood phosphorus and calcium metabolism ; Change in calciuria mmol/d ;Change in urinary pH, urinary specific gravity (g/mL) and crystalluria

SECONDARY OUTCOMES:
Change in volemic parameter | 1 month after initiation of KAFTRIO
  body mass index (BMI) (kg/m²), systolic and diastolic blood pressure (mmHg), presence of orthostatic hypotension, renin and aldosterone levels and ratio (ng/L and pmol/L respectively), natremia (mmol/L), natriuresis (mmol/d), kalemia (mmol/L), kaliuresis (mmol/d), chloremia (mmol/L), bicarbonatemia (mmol/L), brain natriuretic peptid (ng/L), hemoglobin (g/L) and sodium intake estimated by the dietician and calculated thanks to natriuresis (g/d)
Change in volemic parameter | 7 month after initiation of KAFTRIO
  body mass index (BMI) (kg/m²), systolic and diastolic blood pressure (mmHg), presence of orthostatic hypotension, renin and aldosterone levels and ratio (ng/L and pmol/L respectively), natremia (mmol/L), natriuresis (mmol/d), kalemia (mmol/L), kaliuresis (mmol/d), chloremia (mmol/L), bicarbonatemia (mmol/L), brain natriuretic peptid (ng/L), hemoglobin (g/L) and sodium intake estimated by the dietician and calculated thanks to natriuresis (g/d)
Change in renal function | 1 month after initiation of KAFTRIO
  (measured using creatinine (µmol/L) and cystatin C (mg/L)combined to report 2021 CKD-EPIcreatinineand CKD-EPIcreatinine-cystatin C formulas) and in plasma urea levels (mmol/L).
Change in renal function | 7 month after initiation of KAFTRIO
  (measured using creatinine (µmol/L) and cystatin C (mg/L)combined to report 2021 CKD-EPIcreatinineand CKD-EPIcreatinine-cystatin C formulas) and in plasma urea levels (mmol/L).
Change in urinary sediment | 1 month after initiation of KAFTRIO
  , represented by proteinuria (g/day), albuminuria/creatininuria ratio (mg/g) and urinary beta-2-microglobulin level (mg/day), after collecting 24-hours urine sa
Change in urinary sediment | 7 month after initiation of KAFTRIO
  , represented by proteinuria (g/day), albuminuria/creatininuria ratio (mg/g) and urinary beta-2-microglobulin level (mg/day), after collecting 24-hours urine sa
Change in glycemic profile | 1 month after initiation of KAFTRIO
  (fasting blood glucose level (mmol/L) and glycated hemoglobin (%)) and nutritional profile (albumin and pre-albumin in g/L).
Change in glycemic profile | 7 month after initiation of KAFTRIO
  (fasting blood glucose level (mmol/L) and glycated hemoglobin (%)) and nutritional profile (albumin and pre-albumin in g/L).
Change in lung function | 1 month after initiation of KAFTRIO
  predicted forced expiratory volume in 1 second (FEV1) (%) and peak expiratory flow (%)).
Change in lung function | 7 month after initiation of KAFTRIO
  predicted forced expiratory volume in 1 second (FEV1) (%) and peak expiratory flow (%)).

CONTACTS AND LOCATIONS:
Overall Officials: Etienne NOVEL-CATIN, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France